CLINICAL TRIAL: NCT01546857
Title: The Effect of Gabapentin on Postoperative Pain: a Randomized, Double Blind, Placebo Controlled Trial
Brief Title: Effect of Gabapentin on Orthopedic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No longer able to recruit subjects due to unavailability of orthopedic surgeon.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jean Daniel Eloy, MD, J. Daniel Eloy, MD Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011001012
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Degenerative Arthritis and Postoperative Pain
Keywords: orthopedic pain
MeSH Terms: conditions — Osteoarthritis; Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Placebo one dose in the evening of surgery and post op day #1.
  Interventions: Drug: Placebo
- Gabapentin (Active Comparator): Gabapentin 400mg orally at 9pm on the evening of surgery and first day post operatively
  Interventions: Drug: Gapabentin

INTERVENTIONS:
Drug: Placebo — Normal Saline
  Arms: placebo
Drug: Gapabentin — 400mg orally at 9pm day of surgery and the first evening post operatively.
  Other Names: Neurontin
  Arms: Gabapentin

SUMMARY:
This study is being done to determine if a drug called gabapentin helps in the postoperative management of patients undergoing hip and knee operations. The investigators wish to determine the effect of gabapentin on pain and sleep following surgery. If we can lessen a patient's pain and improve sleep, the patient will be better able to participate in their physical therapy. Gabapentin has already been shown to lessen postoperative pain when given before surgery. In healthy patients, it has also been shown to improve certain aspects of sleep. We hope to identify the effect of the drug, when given after surgery, on patients' pain and sleep.

DETAILED DESCRIPTION:
Recent studies have also supported the use of gabapentin as an adjuvant medication in postoperative pain management. Gabapentin decreased the pain associated with movement in post-mastectomy patients. Gilron et al showed a combination of gabapentin and rofecoxib superior to either medication alone in relieving pain after hysterectomy. Later, Gilron et al showed that adding meloxicam to gabapentin in patients undergoing outpatient laparoscopic surgery provided little additional benefit. Clarke et al demonstrated the decrease in the use of opioids in patients who received preoperative and postoperative gabapentin after total knee arthroplasty. They also noted that optimum timing and dosage of the gabapentin needed to be further elucidated. However, in the same year, Clarke et al also reported that gabapentin provided no benefit after total hip arthroplasty when a robust multimodal analgesic regimen was combined with spinal anesthesia. The side effects of gabapentin include sleepiness, which may be of benefit in the postoperative period. In a meta-analysis, Peng showed a 35 % decrease in total opioid consumption in the first 24 hours postoperatively. However, they did note an increase in sleepiness and dizziness. While a recent investigation did not find a connection between sleep disturbances and postoperative pain, a questionnaire study found that the most common reason for nighttime awakenings was pain, and that analgesia was the most helpful intervention. Gabapentin, a structural analogue to y-aminobutyric acid, has been shown in healthy subjects to increase SWS; maintain a stable REM; and reduce arousals, awakenings, and stage shifts-all of which are features of sleep fragmentation. Gabapentin is currently used to treat epilepsy, diabetic neuropathy, postherpetic neuralgia, as well as restless legs syndrome, and its effect on sleep patterns may attribute to its therapeutic success with these disorders Sleep deviates from the normal sleeping pattern in the postoperative patient. Total sleep time, proportion of REM sleep, and proportion of slow wave sleep (SWS) are all reduced. Sleep postoperatively tends to be highly fragmented with multiple spontaneous awakenings and movement arousals. Most of these changes occur during postoperative days 1 and 2; however, patients also incur a REM sleep rebound in days 3 and 4 that can extend up to a week. Studies have demonstrated that these postoperative sleep disturbances, notably the prolonged REM sleep rebound, may contribute to the development of altered mental function, postoperative episodic hypoxemia, and hemodynamic instability. A recent study even found that postoperative sleep disruptions independently predicted functional limitations three months following surgery in patients who underwent total knee replacement. The pathogenesis of these sleep changes appears to be strongly correlated to the magnitude of the surgery as opposed to the type of anesthesia used. Many specific mediators of surgical stress response have been indicated, including catecholamines, cortisol, and IL-1; however, as REM sleep is controlled by many regions of the brain, disturbances may be due to a global excitatory CNS effect.

Our study will recruit 90 patients between the ages of 18 and 70 who are undergoing total hip arthroplasty, hip fracture repair, or total knee arthroplasty and have been assigned an ASA rating of I-III, who are not pregnant. After Institutional Review Board approval, a written informed consent will be obtained from the patient. The study protocol, use of the Patient Controlled Analgesia (PCA) pump, sleep scale, sedation scale, and visual analogue scale for pain will all be explained. Demographic information will be obtained including age, gender, past medical history, past surgical history, hospitalizations, current medications, allergies, and history of drug and alcohol abuse. In addition, a preoperative sleep history will be obtained using the Pittsburgh Sleep Quality Index (PSQI) [14, 15]. The 50 patients will be randomized into two groups: (1) placebo, (2) gabapentin. An Excel generated randomization schedule will be employed. The dosage of gabapentin administered will be 400mg.

Prior to surgery, all patients will be administered midazolam 1-3mg IV to achieve anxiolysis. They will also receive a lumbar plexus block or a femoral nerve block, depending on the surgery to be done, as this has become the standard of care for orthopedic patients at University Hospital. All patients will receive celecoxib 200 mg po bid for three postoperative days. In the operating room, standard general anesthesia technique will be utilized. Upon extubation, the patient will be transferred to the postanesthesia care unit (PACU), where baseline pain and sedation scores will be obtained using the Visual Acuity Scale (VAS), the Richmond Agitation Sedation Scale (RASS), and Ramsay Sedation Scale (RSS), respectively. All pain scores will be assessed with subjects in the resting position. A continuous infusion of bupivacaine 0.125mg/L will be started at a rate of 10mL/hr and continued to postoperative day 2. An I.V. PCA hydromorphone pump will be initiated and set to deliver a 0.2mg bolus per demand with a 5 minute lockout and no background infusion. All patients will be instructed to maintain their VAS pain score at less than 4 out of 10. If the VAS pain score is 5 or greater at rest on two consecutive pain assessments, the dose of intravenous PCA hydromorphone will be increased to deliver a 0.3mg bolus per demand.

At approximately 9pm on the day of the procedure the first dose of placebo/gabapentin will be given. The gabapentin or placebo treatment will be given once more at 9 pm on postoperative day 1. The surgical team will be asked not to order any additional medication for sleep. The following mornings, on POD1 and POD2, a questionnaire addressing the quality of sleep, hours of sleep, number of awakenings throughout the night, and contributing reasons for these awakenings (pain, noise, urination, temperature discomfort, positional discomfort, for nursing care, or other reasons) will be given. Patients will also be assessed for pain, sedation, as well as the incidence of any side effects, including nausea, vomiting, dizziness, and pruritus. In addition, all patients will begin an as-tolerated weight-bearing rehabilitation program for range of motion, strengthening, balance and ambulation beginning the first day after surgery. Success in completion of the physical therapy goals of being out of bed in a chair by postop day 1 and ambulating by postop day 2 will be determined for each group.

The purpose of this study is to determine if a single dose of gabapentin decrease patients' postoperative pain. The primary endpoint will be opioid consumption; additional assessments will include: subjective sleep scales, pain scores, and patient's ability to reach postoperative rehabilitation goals

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a hip arthroplasty, total knee arthroplasty, hip fracture repair American Society of Anesthesiologist rating I-III as determined by your anesthesiologist

Exclusion Criteria:

* Pregnancy and breast feeding

  * An allergy to any of the drugs to be used in the study (midazolam, Celecoxib, gabapentin, hydromorphone, bupivacaine)
  * History of a sleep disorder (Obstructive sleep apnea or daytime somnolence)
  * History of taking chronic narcotic pain medications or gabapentin
  * History of rheumatoid arthritis, a psychiatric disorder, or diabetes with impaired renal function
  * History of alcohol or illicit drug abuse.
  * History of a kidney or liver problem.
  * Inability or unwilling to use patient-controlled analgesia.
  * Unable to meet the criteria for removal of the endotracheal tube in the Operating Room
  * History of asthma, hives or an allergic type reaction following an aspirin or other NSAIDS drug such as Ibuprofen.
  * History of stroke or heart attack or thrombotic event within the past 3 months
  * Lactose intolerance
  * History of cardiac surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Daniel Eloy, MD, Principal Investigator — Rutgers/SUNJ
Locations (1):
- University Hospital, Newark, New Jersey, United States

REFERENCES:
- [Derived] Eloy JD, Anthony C, Amin S, Caparo M, Reilly MC, Shulman S. Gabapentin Does Not Appear to Improve Postoperative Pain and Sleep Patterns in Patients Who Concomitantly Receive Regional Anesthesia for Lower Extremity Orthopedic Surgery: A Randomized Control Trial. Pain Res Manag. 2017;2017:2310382. doi: 10.1155/2017/2310382. Epub 2017 Feb 27. PMID 28348503
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28348503

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo one dose in the evening of surgery and post op day #1.
  Placebo: Placebo
Period: Overall Study
Arm/Group | Placebo | Gabapentin
Started | 14 | 20
Completed | 12 | 17
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Population: we enrolled 34 patients, however 5 subjects withdrew fro the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Categorical [Count of Participants; unit: Participants] — Population: We enrolled 34 subjects but 5 withdrew from the study.
  Participants
    number analyzed (Participants) | 12 | 17 | 29
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 17 | 29
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53.33 [48 to 60] | 54.6 [50 to 64] | 54.1 [48 to 64]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 34 subject were enrolled but 5 withdrew from the study.
  Participants
    number analyzed (Participants) | 12 | 17 | 29
    Female | 6 | 7 | 13
    Male | 6 | 10 | 16
Region of Enrollment [Count of Participants; unit: Participants] — Number of participants
  Participants
    United States | 12 | 17 | 29
ASA Class [Count of Participants; unit: Participants] — Anesthesiology Physical Status for disease severity with ASA 1 classifying healthy subject and ASA 3 specifying more disease severity. Population: 34 subjects were enrolled but 5 withdrew from the study.
  Participants
    number analyzed (Participants) | 12 | 17 | 29
    Class 1 | 0 | 1 | 1
    Class 2 | 5 | 5 | 10
    Class 3 | 7 | 11 | 18
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — PSQI is a self-rating questionnaire used to measure the quality and other parameters of sleep in adults. The PSQI is comprised of seven categories which are graded and equally weighed on a scale from"0" to "3" with the value of "3" being the most negative endpoint. The categories are subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The seven components are added up to a global score which ranges between "0" and "21" with higher scores indicating worse sleep quality. Population: while we enrolled 34 subjects, 5 withdrew from the study.
  units on a scale
    number analyzed (Participants) | 12 | 17 | 29
    (all) | 7.333 (4.355) | 6.765 (3.562) | 7.0 (3.796)

OUTCOME MEASURES:

1. Primary Outcome: Quality of Sleep.
Description: A questionnaire was administered asking participants about the quality of their sleep on the night of surgery asked on postoperative day 1, and on the first postoperative night ( POD 2) . Scored on a scale of zero to 3. Zero meaning poor postoperative sleep and 3 indicating better postoperative sleep.
Time Frame: Night of surgery (POD 1) and Postoperative Day 2.(POD 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 12 | 17
units on a scale
  POD 1 | 1.333 (0.651) | 1.235 (1.091)
  POD 2 | 1 (0.853) | 0.647 (0.862)

2. Primary Outcome: Opioid Consumption
Description: Patient Controlled Analgesia use over 48 hours reported in Morphine equivalent dosage.
Time Frame: 48 hours post operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 12 | 17
mg | 11.88 (6.3) | 11.02 (9.75)

3. Secondary Outcome: Visual Analogue Scale for Pain
Description: Severity of pain measure on a scale from zero to ten. Zero no pain to ten severe pain.
Time Frame: 48 hours post operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 12 | 17
units on a scale | 5.15 (2.28) | 4.38 (3.0)

4. Secondary Outcome: Number of Participants Reaching Rehab Goals.
Time Frame: Duration of hospital stay up to 48 hours
Population: These data were not collected.
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 0/12 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes